CLINICAL TRIAL: NCT00874939
Title: A Randomized Clinical Trial To Evaluate the Single Dose Acute Effects of MK-0249 and Donepezil On Cognitive Function In Adult Patients With Alzheimer's Disease
Brief Title: A Study to Evaluate the Effects of MK-0249 and an Alzheimer's Disease Medication on Cognitive Function in Adults With Alzheimer's Disease (MK-0249-023)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0249-023; MK-0249-023 (Other: Merck Sharp & Dohme Corp.); 2009_572
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — MK-0249; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- PBO→MK-7.5→DON→MK-25 (Experimental): Treatment by single oral dose with Placebo (PBO) in the first crossover period; MK-0249 7.5 mg (MK-7.5) in the second crossover period; Donepezil 5 mg (DON) in the third crossover period; and MK-0249 25 mg (MK-25) in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- MK-7.5→PBO→MK-25→DON (Experimental): Treatment by single oral dose with MK-0249 7.5 mg in the first crossover period; Placebo in the second crossover period; MK-0249 25 mg in the third crossover period; and Donepezil 5 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- DON→MK-25→PBO→MK-7.5 (Experimental): Treatment by single oral dose with Donepezil 5 mg in the first crossover period; MK-0249 25 mg in the second crossover period; Placebo in the third crossover period; and MK-0249 7.5 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- MK-25→DON→MK-7.5→PBO (Experimental): Treatment by single oral dose with MK-0249 25 mg in the first crossover period; Donepezil 5 mg in the second crossover period; MK-0249 7.5 mg in the third crossover period; and Placebo in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- PBO→MK-25→MK-7.5→DON (Experimental): Treatment by single oral dose with Placebo in the first crossover period; MK-0249 25 mg in the second crossover period; MK-0249 7.5 mg in the third crossover period; and Donepezil 5 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- MK-7.5→DON→PBO→MK-25 (Experimental): Treatment by single oral dose with MK-0249 7.5 mg in the first crossover period; Donepezil 5 mg in the second crossover period; Placebo in the third crossover period; and MK-0249 25 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- DON→MK-7.5→MK-25→PBO (Experimental): Treatment by single oral dose with Donepezil 5 mg in the first crossover period; MK-0249 7.5 mg in the second crossover period; MK-0249 25 mg in the third crossover period; and Placebo in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- MK-25→PBO→DON→MK-7.5 (Experimental): Treatment by single oral dose with MK-0249 25 mg in the first crossover period; Placebo in the second crossover period; Donepezil 5 mg in the third crossover period; and MK-0249 7.5 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- PBO→DON→MK-25→MK-7.5 (Experimental): Treatment by single oral dose with Placebo in the first crossover period; Donepezil 5 mg in the second crossover period; MK-0249 25 mg in the third crossover period; and MK-0249 7.5 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- MK-7.5→MK-25→DON→PBO (Experimental): Treatment by single oral dose with MK-0249 7.5 mg in the first crossover period; MK-0249 25 mg in the second crossover period; Donepezil 5 mg in the third crossover period; and Placebo in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- DON→PBO→MK-7.5→MK-25 (Experimental): Treatment by single oral dose with Donepezil 5 mg in the first crossover period; Placebo in the second crossover period; MK-0249 7.5 mg in the third crossover period; and MK-0249 25 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil
- MK-25→MK-7.5→PBO→DON (Experimental): Treatment by single oral dose with MK-0249 25 mg in the first crossover period; MK-0249 7.5 mg in the second crossover period; Placebo in the third crossover period; and Donepezil 5 mg in the fourth crossover period.
  Interventions: Drug: MK-0249 7.5 mg; Drug: MK-0249 25 mg; Drug: Donepezil 5mg; Drug: Placebo to MK-0249; Drug: Placebo to Donepezil

INTERVENTIONS:
Drug: MK-0249 7.5 mg — 4 tablets (1 x 0.5 mg + 2 x 1 mg + 1 x 5 mg) totaling 7.5 mg, single oral dose during each crossover period
Drug: MK-0249 25 mg — 5 x 5 mg tablets totaling 25 mg, single oral dose during each crossover period
Drug: Donepezil 5mg — One 5 mg tablet, single oral dose during each crossover period
  Other Names: Aricept
Drug: Placebo to MK-0249 — Five tablets, single oral dose during each crossover period
Drug: Placebo to Donepezil — One over-encapsulated capsule, single oral dose during each crossover period

SUMMARY:
This study will evaluate acute symptomatic improvements in cognitive performance in healthy elderly participants with mild-to-moderate Alzheimer's disease. A four-week pilot study will first evaluate the CogState computerized cognitive battery in participants who are not receiving treatment. After completion of the pilot study, participants will be randomized to receive Placebo, Donepezil 5 mg, MK-0249 7.5 mg, and MK-0249 25 mg. After each drug administration the participants will be given the CogState computerized cognitive battery to assess cognitive performance. The primary hypotheses are that cognitive performance in participants with Alzheimer's disease, or in healthy participants, is improved by the administration of a single oral 5 mg dose of Donepezil as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Patient Specific:

* Female is not of reproductive potential
* Male who has a female partner(s) of child bearing potential, agrees to use acceptable method of contraception during the study
* Has at least 10 years of education or work history
* Has been a nonsmoker or has not used nicotine for at least 6 months
* Has a diagnosis of mild-to-moderate Alzheimer's Disease
* Has a reliable caregiver who consents to accompany the patient to all clinic visits, provide information to the study staff, and return for follow-up visits and procedures

Healthy Elderly Volunteer Specific:

* Is in good general health
* Has no clinically significant abnormality on electrocardiogram (ECG)

Exclusion Criteria:

Participant Specific:

* Has a history of a neurological disorder other than Alzheimer's disease
* Is living in a nursing home
* Has a history of stroke
* Has a history of psychotic disorder, an active major depressive disorder, or history of schizophrenia
* Has a history of a sleep disorder
* Has a history of a cardiovascular disorder
* Has a history of malignancy
* Is participating or has participated in a study with an investigational compound, device, or vaccine for Alzheimer's disease
* Consumes greater than 6 servings of caffeine (coffee, tea or cola etc.) per day
* Consumes greater than 3 alcoholic beverages per day
* Has had major surgery, donated or loss blood in past 8 weeks

Healthy Elderly Volunteer Specific:

* Is mentally or legally incapacitated, has significant emotional problems, or has a history of a psychiatric disorder over the last 5-10 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-04-06 (Actual); Primary Completion 2009-04-20 (Actual); Study Completion 2009-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight participants were screened and four were enrolled in the study.
Pre-assignment Details: The study was terminated prior to randomization and treatment.
Groups:
- All Participants: All enrolled participants
Period: Overall Study
Arm/Group | All Participants
Started | 4
Treated | 0
Completed | 0
Not Completed | 4
Not completed — Study terminated | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Average of the Change From Baseline After Single Dose Administration of Donepezil 5 mg or Placebo, Measured by Groton Maze Learning Test (GMLT) in Participants With Alzheimer's Disease
Description: The GMLT measures executive function and spatial problem solving on a computer touch screen where participants learn a hidden pathway through a maze consisting of a 10 x 10 grid of tiles. The number of errors made for five consecutive trials at a single session is totaled, where lower number of errors indicates better performance. A change from baseline that is positive indicates improved function.
Time Frame: Baseline and 5-7 hours post-dose
Population: Analysis was not performed due to termination of the study prior to randomization and treatment.
Groups:
- Placebo: Participants treated with Placebo for MK-0249 tablets and Placebo for Donepezil capsule, by single oral dose during each crossover period.
- Donepezil 5 mg: Participants treated with Placebo for MK-0249 tablets, and Donepezil 5 mg capsule, by single oral dose during each crossover period.
Arm/Group | Placebo | Donepezil 5 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time Weighted Average of the Change From Baseline After Single Dose Administration of MK-0249, Measured by GMLT in Participants With Alzheimer's Disease.
Description: as for outcome 1
Time Frame: Baseline and 5-7 hours post-dose
Population: Analysis was not performed due to termination of the study prior to randomization and treatment.
Groups:
- MK-0249 7.5 mg: Participants treated with MK-0249 7.5 mg tablets + a single MK-0249 placebo tablet and Placebo for Donepezil capsule, by single oral dose during each crossover period.
- MK-0249 25 mg: Participants treated with MK-0249 25 mg tablets and Placebo for Donepezil capsule, by single oral dose during each crossover period.
Arm/Group | MK-0249 7.5 mg | MK-0249 25 mg
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Time Weighted Average of the Change From Baseline After Single Dose Administration of Donepezil 5 mg or Placebo, Measured by Groton Maze Learning Test (GMLT) in Healthy Participants
Description: as for outcome 1
Time Frame: Baseline and 5-7 hours post-dose
Population: Analysis was not performed due to termination of the study prior to randomization and treatment.
Arm/Group | Placebo | Donepezil 5 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time Weighted Average of the Change From Baseline After Single Dose Administration of MK-0249, Measured by GMLT in Healthy Participants.
Description: as for outcome 1
Time Frame: Baseline and 5-7 hours post-dose
Population: Analysis was not performed due to termination of the study prior to randomization and treatment.
Arm/Group | MK-0249 7.5 mg | MK-0249 25 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days after last dose of study drug (approximately 67 days)
Description: Participants did not receive any study drug, and therefore were not at risk for adverse events due to termination of the study prior to randomization and treatment.
Arm/Group | MK-0249 7.5 mg | Donepezil 5 mg | MK-0249 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.